CLINICAL TRIAL: NCT05441228
Title: Comparison of Effectiveness of Virtual Reality With Mirror Therapy in Improving Motor Function of Upper Limb of Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shifa Tameer-e-Millat University (Other)
Responsible Party: Principal Investigator, Nouman Khan, Lecturer, Shifa Tameer-e-Millat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Saleha 279-21
Record Dates: First submitted 2022-06-27; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Stroke
Keywords: virtual reallity; Mirror therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: The participant are divided into two groups. The group a received virtual reality and group b received mirror therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A receives virtual reality through Oculus Quest 2. Beat saber application will be used to improve upper limb's motor function of stroke patients. Total 1 hour session will be provided to each patient for 5 days a week. Total period 4 weeks
  Interventions: Device: Oculus Quest 2
- Group B (Other): Group B receives mirror therapy through mirror therapy box. Total 1 hour session will be provided to each patient for 5 days a week. Total period 4 weeks
  Interventions: Device: Mirror therapy box

INTERVENTIONS:
Device: Oculus Quest 2 — Oculus Quest 2 is virtual reality headset with 2 hand control remotes. Beat Saber application will be used on Oculus Quest 2.
  Arms: Group A
Device: Mirror therapy box — Mirror therapy is provided by mirror therapy box by placing it in sagittal plane of patient.
  Arms: Group B

SUMMARY:
The purpose of the study is to compare the effectiveness of virtual reality and mirror therapy in stroke patients. Different studies has been done to find out the best therapy for stroke patients. Use of virtual reality in medical field is becoming more popular now-a-days. Different devices and applications are available to treat various conditions. Research has been done to find the clinical applications of virtual reality for upper limb motor rehabilitation in stroke. in another study, mirror therapy with bilateral arm training was used for hemiplegic upper extremity motor functions in patients with chronic stroke. After doing literature review, it was found that no research has been done to compare the effectiveness of mirror therapy with virtual reality in improving motor function of upper limb of stroke patients. So, In this study these two therapies are compared. For virtual reality Oculus Quest 2 has been used. Patients were allowed to use beat saber game on Oculus.

ELIGIBILITY:
Inclusion Criteria:

* Stroke affecting upper limb

Exclusion Criteria:

* mental problem cognitive problem

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-07-20 (Estimated); Study Completion 2022-07-20 (Estimated)

PRIMARY OUTCOMES:
Fugl- Meyer Upper extremity scale | 4 weeks
  Used to assess motor function of upper limb
Action arm research test | 4 weeks
  To check motor activity of upper limb
Wolf motor function | 4 weeks
  To identify motor activity of upper limb

CONTACTS AND LOCATIONS:
Overall Officials: Saleha Qamar, MSPT*, Principal Investigator — Students
Locations (1):
- Shifa tameer e millat university, Islamabad, Federal, Pakistan

REFERENCES:
- [Background] Laver KE, Lange B, George S, Deutsch JE, Saposnik G, Crotty M. Virtual reality for stroke rehabilitation. Cochrane Database Syst Rev. 2017 Nov 20;11(11):CD008349. doi: 10.1002/14651858.CD008349.pub4. PMID 29156493
- [Background] Erhardsson M, Alt Murphy M, Sunnerhagen KS. Commercial head-mounted display virtual reality for upper extremity rehabilitation in chronic stroke: a single-case design study. J Neuroeng Rehabil. 2020 Nov 23;17(1):154. doi: 10.1186/s12984-020-00788-x. PMID 33228710
- [Background] Thieme H, Mehrholz J, Pohl M, Behrens J, Dohle C. Mirror therapy for improving motor function after stroke. Stroke. 2013 Jan;44(1):e1-2. doi: 10.1161/strokeaha.112.673087. PMID 23390640
- [Background] Dahms C, Brodoehl S, Witte OW, Klingner CM. The importance of different learning stages for motor sequence learning after stroke. Hum Brain Mapp. 2020 Jan;41(1):270-286. doi: 10.1002/hbm.24793. Epub 2019 Sep 14. PMID 31520506
- [Background] Lohse KR, Hilderman CG, Cheung KL, Tatla S, Van der Loos HF. Virtual reality therapy for adults post-stroke: a systematic review and meta-analysis exploring virtual environments and commercial games in therapy. PLoS One. 2014 Mar 28;9(3):e93318. doi: 10.1371/journal.pone.0093318. eCollection 2014. PMID 24681826